CLINICAL TRIAL: NCT04096365
Title: Subcostal Temporary Extracardiac Pacing Study: Clinical Study of the AtaCor Extracardiac Pacing System
Brief Title: Subcostal Temporary Extracardiac Pacing Study
Acronym: STEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AtaCor Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DOC-10052
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Results first posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Conduction Defect
Keywords: Temporary; Ventricular; Pacing
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Subcostal temporary extracardiac pacing lead (Experimental): All subjects will receive a subcostal temporary extracardiac pacing lead for a minimum of 48 hours in-hospital and undergo all protocol testing.
  Interventions: Device: Subcostal Temporary Extracardiac Pacing Lead

INTERVENTIONS:
Device: Subcostal Temporary Extracardiac Pacing Lead — The StealthTrac Lead is designed to facilitate extracardiac temporary ventricular pacing and sensing. The distal end of the StealthTrac Lead is designed to reside within the connective tissue of the anterior mediastinum outside the pericardium. The StealthTrac Lead is delivered using the MACH I Delivery Tool, which is designed to facilitate insertion of the StealthTrac Lead through a small skin incision parallel to the sternum, without the need for fluoroscopic guidance.

SUMMARY:
Up to 15 subjects will be enrolled to evaluate initial safety and performance of the AtaCor Temporary Pacing System. Safety will be evaluated through analysis of all Adverse Events. Performance will be evaluated through (1) the incidence of successful StealthTrac Lead placement using the MACH I Delivery Tool, (2) electrical performance measurements, such as pacing capture thresholds, sensed R-wave amplitudes, pacing impedance and skeletal muscle stimulation at rest. Appropriate sensing and pacing capture will be ascertained from ECG Holter Monitor recordings during periods of in-hospital ambulation.

DETAILED DESCRIPTION:
Enrolled Subjects will have both a market-released transvenous pacing lead and investigational StealthTrac Temporary Pacing Lead placed and evaluated. During the placement procedure, diagnostic echocardiograms will be performed to detect any new pericardial effusions. Once inserted, the StealthTrac Lead will be used to deliver high rate pacing (160 to 220 BPM) in clinically appropriate Subjects, to demonstrate suitability for use in transcatheter procedures that require brief periods of temporary pacing. Lead positions will be documented using fluoroscopic images before the Subject leaves the procedure room. On the following two days after the procedure, electrical performance will be evaluated in multiple postures and appropriate pacing and sensing will be confirmed during activity using ECG Holter monitor recordings. Subjects will also be asked patient-centric questions about their experience with the StealthTrac Lead throughout the study period. Evaluations will continue for a minimum of two (2) and a maximum of seven (7) days after the index procedure. Prior to StealthTrac Lead removal, an X-Ray will be taken to document the final lead position and diagnostic echocardiography will be performed to (1) detect any latent pericardial effusions and (2) assess differences in cardiac function with intrinsic conduction and while pacing. A final follow-up will be performed 25-30 days after removal to identify any latent adverse events before the Subject exits the study.

ELIGIBILITY:
Inclusion Criteria:

1. Indicated for closed-chest cardiac invasive procedure with the potential for intra-procedural or post-procedural bradycardia and willing to be hospitalized for a minimum of 2 days post procedure.

   Examples of such procedures include: transfemoral transcatheter aortic valve replacement (TAVR), balloon valvuloplasty, permanent pacemaker implantation and pacing lead extractions/revisions.
2. Physically and mentally capable of providing informed consent.
3. At least 18 years of age or of legal age to provide consent as required by local and national requirements.

Exclusion Criteria:

1. Contraindicated or clinically unsuitable for transvenous lead placement;
2. Implanted with an implantable cardioverter defibrillator (ICD) or transvenous defibrillation lead at the time of enrollment;
3. History of a prior sternotomy (median or partial);
4. History of prior surgery with disruption of the lung, pericardium or connective tissue between the sternum and pericardium;
5. History of significant anatomic derangement of the thorax (e.g., pectus excavatum), prior chest radiation therapy or other reasons which may cause pericardial adhesions or complicate the AtaCor Temporary Pacing System insertion procedure;
6. History of pericardial disease, pericarditis or mediastinitis;
7. History of chronic obstructive pulmonary disease (COPD);
8. NYHA functional classification IV at the time of enrollment;
9. History of congenital heart disease;
10. Patients with circumstances that prevent data collection or follow-up, including conditions that prevent ambulation and testing in multiple postures;
11. BMI ≥ 35 kg/m2;
12. History of allergies to any study device components;
13. Pregnant or lactating (current or anticipated during study follow up); and
14. Participation in any concurrent study without prior, written approval from the Sponsor.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-08-25 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2019-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Burke, D.O., Principal Investigator — AtaCor Medical; Adrian Ebner, M.D., Principal Investigator — Sanatorio Italiano
Locations (1):
- Sanatorio Italiano, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor website — https://www.atacor.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eleven (11) of the 12 enrolled subjects underwent a StealthTrac Lead insertion procedure. One (1) subject experienced an adverse clinical event, unrelated to the StealthTrac Lead, that precluded insertion of the StealthTrac Lead and was subsequently withdrawn from the study.
Period: Overall Study
Arm/Group | Subcostal Temporary Extracardiac Pacing Lead
Started | 12
Completed | 11
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Subcostal Temporary Extracardiac Pacing Lead
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Mestizo / Indigenous | 6
  White / Caucasian | 5
Region of Enrollment [Number; unit: participants]
  Paraguay | 11

OUTCOME MEASURES:

1. Primary Outcome: Safety Outcome: Number of Subjects Experiencing an Adverse Device Effect
Description: Safety will be evaluated through analysis of all Adverse Device Effects
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Subcostal Temporary Extracardiac Pacing Lead
Number analyzed (Participants) | 11
Participants | 2

2. Primary Outcome: Performance Outcome: Mean Pacing Capture Threshold (V)
Description: Minimum current required to pacing the heart (in multiple postures)
Time Frame: Up to 2 days post insertion
Population: One suspected lead dislodgement prevented measurements in all 11 subjects on Day 1 and Day 2.
Measure: Mean (Standard Deviation); unit: Volts
Arm/Group | Subcostal Temporary Extracardiac Pacing Lead
Number analyzed (Participants) | 11
Volts
  Day 0 (Procedure) | 4.1 (1.4)
  Day 1: number analyzed (Participants) | 10
  Day 1 | 5.6 (2.7)
  Day 2: number analyzed (Participants) | 10
  Day 2 | 7.0 (2.6)

3. Primary Outcome: Performance Outcome: Mean Pacing Impedance (Ohms)
Description: Impedance measured while pacing the heart (in multiple postures)
Time Frame: Up to 2 days post insertion
Population: All eleven (11) Subjects contribute data on Day 0. On Day 1 and Day 2, nine (9) Subjects contribute data and two (2) Subjects do not due to a suspected lead dislodgement and one measurement out of range.
Measure: Mean (Standard Deviation); unit: Ohms
Arm/Group | Subcostal Temporary Extracardiac Pacing Lead
Number analyzed (Participants) | 11
Ohms
  Day 0 | 557 (176)
  Day 1: number analyzed (Participants) | 9
  Day 1 | 320 (115)
  Day 2: number analyzed (Participants) | 9
  Day 2 | 266 (60)

4. Primary Outcome: Performance Outcome: Mean R-Wave Amplitude (mV)
Description: R-Wave amplitudes measured while sensing the heart (in multiple postures)
Time Frame: Up to 2 days post insertion
Population: Only 4 of 11 subjects had an intrinsic rhythm for measurement of R waves.
Measure: Mean (Standard Deviation); unit: millivolts
Arm/Group | Subcostal Temporary Extracardiac Pacing Lead
Number analyzed (Participants) | 4
millivolts
  Day 0 | 4.9 (1.7)
  Day 1 | 2.7 (1.3)
  Day 2 | 2.6 (1.4)

5. Primary Outcome: Performance Outcome: % of R-R Intervals With Appropriate Pacing and Sensing During Activity
Description: ECG Holter Recordings obtained during periods of rest and in-hospital activity. The % of R-R intervals with appropriate pacing is calculated as the number of paced intervals that demonstrate pacing capture / the total number of pacing intervals. The % of R-R intervals with appropriate sensing is calculated as the number of intervals where pacing is appropriately delivered or inhibited (depending on the programmed settings of the pacemaker) / the total number of R-R intervals. The outcomes are presented a % of intervals and not an average of the percentages observed across patients.
Time Frame: Up to 2 days post insertion
Population: All subjects with a StealthTrac Lead
Measure: Number; unit: % of intervals
Arm/Group | Subcostal Temporary Extracardiac Pacing Lead
Number analyzed (Participants) | 11
% of intervals
  Pacing Capture | 97.85
  Appropriate Sensing | 98.9

6. Other Pre Specified Outcome: Paced QRS Duration (ms)
Description: QRS duration measured from 12-Lead ECG
Time Frame: 1 day after insertion
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Echocardiographic Assessment of Left Ventricular Stroke Volume During Pacing (mL)
Description: Measures of cardiac function obtained from echocardiography
Time Frame: 2 days after insertion
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 Days
Arm/Group | Subcostal Temporary Extracardiac Pacing Lead
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 2/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subcostal Temporary Extracardiac Pacing Lead (N=11)
Pain (Post-Operative) (Surgical and medical procedures) | 2 (2)
Inability to Pace (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator must obtain prior written consent of Sponsor before publishing.

DOCUMENTS (1):
  • Study Protocol (2019-07-23): https://cdn.clinicaltrials.gov/large-docs/65/NCT04096365/Prot_001.pdf